CLINICAL TRIAL: NCT03690388
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Cabozantinib (XL184) in Subjects With Radioiodine-Refractory Differentiated Thyroid Cancer Who Have Progressed After Prior Vascular Endothelial Growth Factor Receptor (VEGFR) -Targeted Therapy
Brief Title: A Study of Cabozantinib Compared With Placebo in Subjects With Radioiodine-refractory Differentiated Thyroid Cancer Who Have Progressed After Prior Vascular Endothelial Growth Factor Receptor (VEGFR) -Targeted Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XL184-311; 2024-516478-31-00 (EU CTIS Number)
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Thyroid cancer, papillary; Papillary thyroid carcinoma; Nonmedullary thyroid carcinoma; Cancer of the thyroid; Thyroid cancer; Follicular thyroid cancer; Thyroid cancer, follicular; Hürthle cell cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid cancer, follicular | interventions — cabozantinib

STUDY DESIGN:
Intervention Model Description: This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study of cabozantinib in subjects with radioactive iodine (RAI)-refractory differentiated thyroid cancer (DTC) after prior vascular endothelial growth factor receptor (VEGFR)-tyrosine kinase inhibitor (TKI) therapy. Cabozantinib-matched placebo will be given in the control arm to blind (mask) study treatment. Approximately 300 eligible subjects will be randomized in a 2:1 ratio to receive either cabozantinib or placebo. After the primary efficacy endpoints have been analyzed and sufficient data have been collected to adequately evaluate all study endpoints to establish, for regulatory purposes, the safety and efficacy profile of the experimental drug within this study, the study will transition to an open label Maintenance Phase.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study treatment assignment will be unknown to the subjects, investigators, study centers, Sponsor, and any Contract Research Organization affiliated with the study other than those authorized to access treatment assignment for regulatory safety reporting and submission processes, interactive response technology (IRT) system administration, and drug supply management. Cabozantinib-matched placebo will be packaged and color-, size-, and shape-matched to be indistinguishable from cabozantinib. Individual study treatment assignment will be unblinded and information provided to the Investigators upon request for subjects with radiographic progressive disease (PD) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 confirmed by the blinded independent radiology committee (BIRC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cabozantinib (Experimental): cabozantinib (60 mg) once daily orally (qd)
  Interventions: Drug: Cabozantinib
- Placebo (Placebo Comparator): placebo once daily orally (qd)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabozantinib — Tablets containing 60-mg or 20-mg cabozantinib once daily orally.
  Other Names: XL184; Cabometyx®
  Arms: Cabozantinib
Drug: Placebo — Tablets containing placebo equivalent of 60-mg or 20-mg cabozantinib once daily orally.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the effect of cabozantinib compared with placebo on progression free survival (PFS) and objective response rate (ORR) in subjects with Radioiodine-Refractory Differentiated Thyroid Cancer (DTC) who have progressed after prior vascular endothelial growth factor receptor (VEGFR)-Targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of Differentiated Thyroid Cancer (DTC)
2. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
3. Previously treated with or deemed ineligible for treatment with Iodine- 131 for differentiated thyroid cancer (DTC)
4. Previously treated with at least one of the following vascular endothelial growth factor receptor (VEGFR)-targeting tyrosine kinase inhibitor (TKI) agents for DTC: lenvatinib or sorafenib. Note: Up to two prior VEGFR-targeting TKI agents are allowed
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1

Exclusion Criteria:

1. Prior treatment with any of the following: Cabozantinib; Selective small-molecule v-raf murine sarcoma viral oncogene homolog B1 (BRAF) kinase inhibitor; More than 2 VEGFR-targeting TKI agents; More than 1 immune checkpoint inhibitor therapy; 1 systemic chemotherapy regimen (given as single agent or in combination with another chemotherapy agent)
2. Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks or 5 half-lives of the agent, whichever is longer, before randomization
3. Receipt of any type of anticancer antibody (including investigational antibody) or systemic chemotherapy within 4 weeks before randomization
4. Receipt of radiation therapy for bone metastasis within 2 weeks or any other radiation therapy within 4 weeks before randomization.
5. Known brain metastases or cranial epidural disease unless adequately treated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (164):
- United States (31):
  - Exelixis Clinical Site #2, Newport Beach, California
  - Exelixis Clinical Site #98, Sacramento, California
  - Exelixis Clinical Site #69, San Francisco, California
  - Exelixis Clinical Site #10, Stanford, California
  - Exelixis Clinical Site #3, Torrance, California
  - Exelixis Clinical Site #9, Aurora, Colorado
  - Exelixis Clinical Site #21, New Haven, Connecticut
  - Exelixis Clinical Site #4, Washington D.C., District of Columbia
  - Exelixis Clinical Site #94, Miami, Florida
  - Exelixis Clinical Site #93, Orlando, Florida
  - Exelixis Clinical Site #6, Tampa, Florida
  - Exelixis Clinical Site #164, Chicago, Illinois
  - Exelixis Clinical Site #54, Lexington, Kentucky
  - Exelixis Clinical Site #153, Boston, Massachusetts
  - Exelixis Clinical Site #80, Ann Arbor, Michigan
  - Exelixis Clinical Site #78, Detroit, Michigan
  - Exelixis Clinical Site #22, Detroit, Michigan
  - Exelixis Clinical Site #63, Columbia, Missouri
  - Exelixis Clinical Site #42, St Louis, Missouri
  - Exelixis Clinical Site #11, Omaha, Nebraska
  - Exelixis Clinical Site #118, Morristown, New Jersey
  - Exelixis Clinical Site #76, Charlotte, North Carolina
  - Exelixis Clinical Site #19, Durham, North Carolina
  - Exelixis Clinical Site #7, Cincinnati, Ohio
  - Exelixis Clinical Site #5, Bethlehem, Pennsylvania
  - Exelixis Clinical Site #1, Philadelphia, Pennsylvania
  - Exelixis Clinical Site #75, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #134, Charleston, South Carolina
  - Exelixis Clinical Site #68, Nashville, Tennessee
  - Exelixis Clinical Site #8, Houston, Texas
  - Exelixis Clinical Site #113, Seattle, Washington
- Argentina (3):
  - Exelixis Clinical Site #96, Pergamino, Buenos Aires
  - Exelixis Clinical Site #97, Caba
  - Exelixis Clinical Site #129, Córdoba
- Australia (5):
  - Exelixis Clinical Site #17, St Leonards, New South Wales
  - Exelixis Clinical Site #25, Waratah, New South Wales
  - Exelixis Clinical Site #86, Bedford Park, South Australia
  - Exelixis Clinical Site #24, Melbourne, Victoria
  - Exelixis Clinical Site #12, Herston
- Austria (2):
  - Exelixis Clinical Site #62, Salzburg
  - Exelixis Clinical Site #119, Vienna
- Belgium (6):
  - Exelixis Clinical Site #90, Anderlecht
  - Exelixis Clinical Site #31, Brussels
  - Exelixis Clinical Site #26, Edegem
  - Exelixis Clinical Site #74, Edegem
  - Exelixis Clinical Site #100, Ghent
  - Exelixis Clinical Site #27, Namur
- Brazil (8):
  - Exelixis Clinical Site #35, Cascavel, Paraná
  - Exelixis Clinical Site #39, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #140, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #38, Porto Alegre, Rio Grande do Sul
  - Exelixis Clinical Site #116, Ribeirão Preto, São Paulo
  - Exelixis Clinical Site #40, São José do Rio Preto, São Paulo
  - Exelixis Clinical Site #92, Rio de Janeiro
  - Exelixis Clinical Site #47, São Paulo
- Canada (4):
  - Exelixis Clinical Site #20, Calgary, Alberta
  - Exelixis Clinical Site #18, Edmonton, Alberta
  - Exelixis Clinical Site #107, London, Ontario
  - Exelixis Clinical Site #83, Toronto, Ontario
- Croatia (3):
  - Exelixis Clinical Site #145, Osijek
  - Exelixis Clinical Site #137, Zagreb
  - Exelixis Clinical Site #138, Zagreb
- Czechia (2):
  - Exelixis Clinical Site #105, Brno
  - Exelixis Clinical Site #104, Olomouc
- France (10):
  - Exelixis Clinical Site #32, Dijon, Bourgogne-Franche-Comté
  - Exelixis Clinical Site #67, Bordeaux, Nouvelle-Aquitaine
  - Exelixis Clinical Site #45, Angers, Pays de la Loire Region
  - Exelixis Clinical Site #72, Marseille, Provence-Alpes-Côte d'Azur Region
  - Exelixis Clinical Site #102, Besançon
  - Exelixis Clinical Site #91, Lyon
  - Exelixis Clinical Site #82, Nice
  - Exelixis Clinical Site #152, Paris
  - Exelixis Clinical Site #95, Strasbourg
  - Exelixis Clinical Site #44, Villejuif, Île-de-France Region
- Germany (12):
  - Exelixis Clinical Site #121, Tübingen, Baden-Wurttemberg
  - Exelixis Clinical Site #156, Würzburg, Bavaria
  - Exelixis Clinical Site #125, Marburg, Hesse
  - Exelixis Clinical Site #163, Hanover, Lower Saxony
  - Exelixis Clinical Site #151, Dresden, Saxony
  - Exelixis Clinical Site #124, Magdeburg, Saxony-Anhalt
  - Exelixis Clinical Site #155, Aachen
  - Exelixis Clinical Site #131, Bonn
  - Exelixis Clinical Site #154, Essen
  - Exelixis Clinical Site #160, Freiburg im Breisgau
  - Exelixis Clinical Site #159, Hamburg
  - Exelixis Clinical Site #139, München
- Exelixis Clinical Site #28, Hong Kong, Hong Kong
- Hungary (2):
  - Exelixis Clinical Site #46, Budapest
  - Exelixis Clinical Site #37, Pécs
- Israel (3):
  - Exelixis Clinical Site #43, Haifa
  - Exelixis Clinical Site #41, Jerusalem
  - Exelixis Clinical Site #58, Petah Tikva
- Italy (16):
  - Exelixis Clinical Site #109, Viagrande, Catania
  - Exelixis Clinical Site #135, Catania, CT
  - Exelixis Clinical Site #132, Meldola, Forlì - Cesena
  - Exelixis Clinical Site #144, Genova, GE
  - Exelixis Clinical Site #143, Rozzano, Milano
  - Exelixis Clinical Site #29, Pisa, PI
  - Exelixis Clinical Site #120, Torino, TO
  - Exelixis Clinical Site #103, Milan
  - Exelixis Clinical Site #110, Milan
  - Exelixis Clinical Site #115, Milan
  - Exelixis Clinical Site #108, Napoli
  - Exelixis Clinical Site #56, Napoli
  - Exelixis Clinical Site #123, Padua
  - Exelixis Clinical Site #87, Roma
  - Exelixis Clinical Site #127, Roma
  - Exelixis Clinical Site #111, Siena
- Mexico (5):
  - Exelixis Clinical Site #158, Tuxtla Gutiérrez, Chiapas
  - Exelixis Clinical Site #133, Ciudad de Mèxico
  - Exelixis Clinical Site #147, Mexico City
  - Exelixis Clinical Site #148, Mexico City
  - Exelixis Clinical Site #161, San Luis Potosí City
- Netherlands (2):
  - Exelixis Clinical Site #128, Amsterdam, North Holland
  - Exelixis Clinical Site #117, Leiden, South Holland
- Poland (3):
  - Exelixis Clinical Site #59, Poznan, Greater Poland Voivodeship
  - Exelixis Clinical Site #15, Warsaw, Masovian Voivodeship
  - Exelixis Clinical Site #61, Gliwice, Silesian Voivodeship
- Romania (4):
  - Exelixis Clinical Site #149, Cluj-Napoca, Cluj
  - Exelixis Clinical Site #150, Craiova, Dolj
  - Exelixis Clinical Site #142, Timișoara, Timiș County
  - Exelixis Clinical Site #146, Bucharest
- Russia (11):
  - Exelixis Clinical Site #48, Obninsk, Kaluzhiskiy Region
  - Exelixis Clinical Site #55, Kislino, Kursk Oblast
  - Exelixis Clinical Site #157, Tyumen, Tyumen Oblast
  - Exelixis Clinical Site #49, Moscow
  - Exelixis Clinical Site #53, Moscow
  - Exelixis Clinical Site #84, Moscow
  - Exelixis Clinical Site #85, Moscow
  - Exelixis Clinical Site #106, Omsk
  - Exelixis Clinical Site #89, Saint Petersburg
  - Exelixis Clinical Site #52, Samara
  - Exelixis Clinical Site #66, Yaroslavl
- South Korea (4):
  - Exelixis Clinical Site #70, Busan
  - Exelixis Clinical Site #79, Gyeonggi-do
  - Exelixis Clinical Site #36, Seoul
  - Exelixis Clinical Site #34, Seoul
- Spain (10):
  - Exelixis Clinical Site #14, Barcelona
  - Exelixis Clinical Site #99, Barcelona
  - Exelixis Clinical Site #114, Madrid
  - Exelixis Clinical Site #30, Madrid
  - Exelixis Clinical Site #13, Madrid
  - Exelixis Clinical Site #16, Madrid
  - Exelixis Clinical Site #33, Madrid
  - Exelixis Clinical Site #73, Madrid
  - Exelixis Clinical Site #23, Madrid
  - Exelixis Clinical Site #81, Málaga
- Taiwan (4):
  - Exelixis Clinical Site #136, Tainan
  - Exelixis Clinical Site #112, Tainan
  - Exelixis Clinical Site #77, Taipei
  - Exelixis Clinical Site #101, Taipei
- Thailand (4):
  - Exelixis Clinical Site #126, Bangkok Noi, Bangkok
  - Exelixis Clinical Site #122, Pathum Wan, Bangkok
  - Exelixis Clinical Site #141, Ratchathewi, Bangkok
  - Exelixis Clinical Site #130, Hat Yai, Changwat Songkhla
- United Kingdom (9):
  - Exelixis Clinical Site #88, Birmingham, England
  - Exelixis Clinical Site #71, Bristol, England
  - Exelixis Clinical Site #162, London, England
  - Exelixis Clinical Site #51, Oxford, England
  - Exelixis Clinical Site #64, Aberdeen, Scotland
  - Exelixis Clinical Site #50, Glasgow, Scotland
  - Exelixis Clinical Site #60, Cardiff, Wales
  - Exelixis Clinical Site #65, Manchester
  - Exelixis Clinical Site #57, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capdevila J, Krajewska J, Hernando J, Robinson B, Sherman SI, Jarzab B, Lin CC, Vaisman F, Hoff AO, Hitre E, Bowles DW, Williamson D, Levytskyy R, Oliver J, Keam B, Brose MS. Increased Progression-Free Survival with Cabozantinib Versus Placebo in Patients with Radioiodine-Refractory Differentiated Thyroid Cancer Irrespective of Prior Vascular Endothelial Growth Factor Receptor-Targeted Therapy and Tumor Histology: A Subgroup Analysis of the COSMIC-311 Study. Thyroid. 2024 Mar;34(3):347-359. doi: 10.1089/thy.2023.0463. Epub 2024 Jan 23. PMID 38062732
- [Derived] Brose MS, Robinson B, Sherman SI, Krajewska J, Lin CC, Vaisman F, Hoff AO, Hitre E, Bowles DW, Hernando J, Faoro L, Banerjee K, Oliver JW, Keam B, Capdevila J. Cabozantinib for radioiodine-refractory differentiated thyroid cancer (COSMIC-311): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1126-1138. doi: 10.1016/S1470-2045(21)00332-6. Epub 2021 Jul 5. PMID 34237250

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib | Placebo
Started | 125 | 62
Completed | 89 | 26
Not Completed | 36 | 36
Not completed — Adverse Event | 8 | 1
Not completed — Radiographic Progression | 14 | 29
Not completed — Clinical deterioration | 10 | 6
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib | Placebo | Total
Number analyzed (Participants) | 125 | 62 | 187
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 29 | 91
  >=65 years | 63 | 33 | 96
Age, Continuous [Median (Full Range); unit: years] | 65 [32 to 85] | 66 [37 to 81] | 66 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 34 | 102
  Male | 57 | 28 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 6 | 27
  Not Hispanic or Latino | 95 | 53 | 148
  Unknown or Not Reported | 9 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 20 | 14 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 90 | 41 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 5 | 16
Region of Enrollment [Number; unit: participants]
  Hong Kong | 0 | 1 | 1
  United States | 10 | 9 | 19
  Czechia | 1 | 0 | 1
  Thailand | 2 | 1 | 3
  Russia | 8 | 3 | 11
  Austria | 4 | 0 | 4
  Netherlands | 1 | 1 | 2
  South Korea | 8 | 8 | 16
  Brazil | 11 | 4 | 15
  Poland | 9 | 4 | 13
  France | 8 | 3 | 11
  Croatia | 1 | 0 | 1
  Argentina | 1 | 0 | 1
  Romania | 3 | 1 | 4
  Hungary | 5 | 3 | 8
  United Kingdom | 4 | 3 | 7
  Spain | 10 | 9 | 19
  Canada | 3 | 0 | 3
  Belgium | 3 | 2 | 5
  Taiwan | 6 | 3 | 9
  Italy | 14 | 5 | 19
  Mexico | 3 | 0 | 3
  Israel | 3 | 0 | 3
  Australia | 5 | 1 | 6
  Germany | 2 | 1 | 3
Receipt of prior lenvatinib [Count of Participants; unit: Participants] | 79 | 39 | 118

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time to the earlier of either radiographic progressive disease (PD) or death from any cause.
Time Frame: Up to approximately twenty months after the first subject is randomized. Time from randomization to the earlier of the following events: radiographic PD as determined by the blinded independent central review (BIRC) or death due to any cause.
Population: All subjects randomized at the time of the analysis (N=187).
Measure: Median (96% Confidence Interval); unit: months
Arm/Group | Cabozantinib | Placebo
Number analyzed (Participants) | 125 | 62
months | NA [5.7 to NA] — The CI 5.7 to 0.0 is not 0.0 but NA. The median PFS and upper bound of the CI could not be determined because not enough subjects on the cabozantinib arm had experienced progression at the time of the data cut-off to determine a median PFS. However, it was possible to estimate the HR at that timepoint based on the Cox Proportional Hazards Model. | 1.9 [1.8 to 3.6]
Statistical Analysis 1: Comparison: Cabozantinib vs Placebo; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.22, 96% CI 2-sided [0.13 to 0.36]

2. Primary Outcome: Objective Response Rate (ORR)
Description: Proportion of subjects with the best overall response of complete response (CR) or partial response (PR).
Time Frame: Six months after 100 subjects are randomized. Time from randomization to best overall response of confirmed complete response (CR) or confirmed partial response (PR) per BIRC per RECIST 1.1.
Population: The first 100 subjects randomized.
Measure: Number (99% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib | Placebo
Number analyzed (Participants) | 67 | 33
percentage of participants | 15 [5.8 to 29.3] | 0 [0.0 to 14.8]

ADVERSE EVENTS:
Time Frame: 1 year, 8 months.
Description: Safety assessments included evaluations of AEs, SAEs, deaths, clinical laboratory test results (hematology, serum chemistry, and urinalysis), physical examination findings, vital sign measurements, Eastern Cooperative Oncology Group performance status (ECOG PS), and 12-lead ECG recordings.
Arm/Group | Cabozantinib | Placebo
All-Cause Mortality (participants affected / at risk) | 17/125 | 14/62
Serious Adverse Events (participants affected / at risk) | 43/125 | 18/62
Other Adverse Events (participants affected / at risk) | 112/125 | 32/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=125) | Placebo (N=62)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Anal abscess (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=125) | Placebo (N=62)
Diarrhoea (Gastrointestinal disorders) | 69 | 2
Nausea (Gastrointestinal disorders) | 33 | 1
Vomiting (Gastrointestinal disorders) | 18 | 5
Stomatitis (Gastrointestinal disorders) | 20 | 2
Constipation (Gastrointestinal disorders) | 14 | 5
Dry mouth (Gastrointestinal disorders) | 13 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 2
Dyspepsia (Gastrointestinal disorders) | 7 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 59 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 1
Fatigue (General disorders) | 41 | 5
Asthenia (General disorders) | 21 | 9
Mucosal inflammation (General disorders) | 18 | 0
Decreased appetite (Metabolism and nutrition disorders) | 33 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 30 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 1
Alanine aminotransferase increased (Investigations) | 32 | 1
Aspartate aminotransferase increased (Investigations) | 32 | 1
Weight decreased (Investigations) | 25 | 3
Blood lactate dehydrogenase increased (Investigations) | 12 | 0
Blood alkaline phosphatase increased (Investigations) | 13 | 2
Neutrophil count decreased (Investigations) | 7 | 1
Platelet count decreased (Investigations) | 8 | 1
Hypertension (Vascular disorders) | 37 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 9
Dysgeusia (Nervous system disorders) | 14 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Headache (Nervous system disorders) | 14 | 1
Proteinuria (Renal and urinary disorders) | 21 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 8
Urinary tract infection (Infections and infestations) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤ 60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03690388/Prot_SAP_000.pdf